CLINICAL TRIAL: NCT01678898
Title: A Phase 1/2, Open Label, Dose Ranging Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Exploratory Efficacy Parameters of PRX-102 Administered by Intravenous Infusion Every 2 Weeks for 12 Months to Adult Fabry Patients
Brief Title: Dose-ranging Study of PRX-102 in Adult Fabry Disease Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Protalix (Industry)
Collaborators: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PB-102-F01 & PB-102-F02; NCT01769001 (obsolete NCT alias)
Record Dates: First submitted 2012-08-31; First posted 2012-09-05 (Estimated); Results first posted 2020-01-27 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Fabry Disease
Keywords: Fabry disease; Alpha galactosidase deficiency; Metabolic storage disease
MeSH Terms: conditions — Fabry Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 0.2 mg/kg (Experimental): PRX-102 0.2 mg/kg every 2 weeks
  Interventions: Drug: PRX-102
- 1 mg/kg (Experimental): PRX-102 1 mg/kg every 2 weeks
  Interventions: Drug: PRX-102
- 2 mg/kg (Experimental): PRX-102 2 mg/kg every 2 weeks
  Interventions: Drug: PRX-102

INTERVENTIONS:
Drug: PRX-102
  Other Names: plant cell expressed recombinant human alpha-galactosidase-A

SUMMARY:
This is the first human treatment with PRX-102, an enzyme being developed as a long-term enzyme replacement therapy in patients with a confirmed diagnosis of Fabry disease (alpha galactosidase deficiency). The safety, tolerability, and exploratory efficacy will be evaluated in this study of increasing doses. Patients will be treated with infusions every two weeks for 12 months.

DETAILED DESCRIPTION:
Under the PB-102-F01 study protocol, patients will be enrolled into one of three PRX-102 dosing groups (0.2 mg/kg, 1.0 mg/kg, 2.0 mg/kg) and receive PRX-102 as an intravenous infusion every 2 weeks for 12 weeks (3 months). Patients who finish the PB-102-F01 study will be enrolled in the PB-102-F02 extension study and receive the same dose they had received in the PB-102-F01 study for an additional 38 weeks (9 months).

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic adult Fabry patients (≥18 yrs)
* Males: plasma and/or leucocyte alpha galactosidase activity (by activity assay) less than lower limit of normal (LLN in plasma=3.2 nmol/hr/ml, LLN in leucocytes=32 nmol/hr/mg/protein)
* Females: historical genetic test results consistent with Fabry mutations
* Globotriaosylceramide (Gb3) concentration in urine > 1.5 times upper normal limit
* Patients who have never received enzyme replacement therapy (ERT) in the past, or patients who have not received ERT in the past 6 months and have a negative anti alpha galactosidase antibody test
* eGFR ≥ 60 mL/min/1.73m2
* The patient signs informed consent
* Female patients and male patients whose co-partners are of child-bearing potential agree to use a medically acceptable method of contraception, not including the rhythm method

Exclusion Criteria:

* Participation in any trial of an investigational drug within 30 days prior to study screening
* Chronic kidney disease stages 3-5 (CKD 3-5) (Appendix 7)
* History of dialysis or renal transplantation
* Angiotensin converting enzyme (ACE) inhibitor or angiotensin receptor blocker (ARB) therapy initiated or dose changed in the 4 weeks prior to screening
* Severe myocardial fibrosis by MRI (≥2 late-enhancement [LE] positive left ventricular segments) (Weidemann et al. 2009)
* History of clinical stroke
* Pregnant or nursing
* Presence of HIV and/or HBsAg and/or Hepatitis C infections
* Known allergies to ERT
* Known allergy to Gadolinium based contrast agents
* Presence of any medical, emotional, behavioral or psychological condition that, in the judgment of the Investigator and/or Medical Director, would interfere with the patient's compliance with the requirements of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2012-10 (Actual); Primary Completion 2016-03-06 (Actual); Study Completion 2016-03-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (14):
- United States (9):
  - UC Davis Medical Center, MIND Institute Department of Pediatrics, Section of Genetics, Sacramento, California
  - Department of Human Genetics, Emory University School of Medicine, Atlanta, Georgia
  - University of Iowa Health Clinics, Iowa City, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - Johns Hopkins University School of Medicine, Baltimore, Maryland
  - Duke University Medical Center, Durham, North Carolina
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Research Baylor Institute of Metabolic Disease, Dallas, Texas
  - O & O Alpan LLC, Fairfax, Virginia
- Royal Melbourne Hospital, Victoria Park, Australia
- Hematology and Clinical Research Private Institute, Asunción, Paraguay
- Clinical Center of Serbia, Belgrade, Serbia
- Hospital de Dia Quiron Zaragoza, Zaragoza, Spain
- The Royal Free Hospital, London, United Kingdom

REFERENCES:
- [Result] Schiffmann R, Goker-Alpan O, Holida M, Giraldo P, Barisoni L, Colvin RB, Jennette CJ, Maegawa G, Boyadjiev SA, Gonzalez D, Nicholls K, Tuffaha A, Atta MG, Rup B, Charney MR, Paz A, Szlaifer M, Alon S, Brill-Almon E, Chertkoff R, Hughes D. Pegunigalsidase alfa, a novel PEGylated enzyme replacement therapy for Fabry disease, provides sustained plasma concentrations and favorable pharmacodynamics: A 1-year Phase 1/2 clinical trial. J Inherit Metab Dis. 2019 May;42(3):534-544. doi: 10.1002/jimd.12080. Epub 2019 Apr 8. PMID 30834538

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment efforts were conducted in North and South America, Europe and Australia for PB-102-F01 (3 months), and all patients who completed this study continued to the PB-102-F02 extension study for an additional 9 months, to complete a total of 12 months of treatment. 18 patients were eligible for enrollment, and 16 completed the study.
Pre-assignment Details: Eighteen (18) patients were eligible for enrollment for PB-102-F01 study. The eligible patients who completed PB-102-F01, needed to sign an informed consent for PB-102-F02.
Groups:
- 0.2 mg/kg: PRX-102 0.2 mg/kg every 2 weeks
  PRX-102
- 1 mg/kg: PRX-102 1 mg/kg every 2 weeks
  PRX-102
- 2 mg/kg: PRX-102 2 mg/kg every 2 weeks
  PRX-102
Period: PB-102-F01
Arm/Group | 0.2 mg/kg | 1 mg/kg | 2 mg/kg
Started | 6 | 8 | 4
Completed | 6 | 6 | 4
Not Completed | 0 | 2 | 0
Not completed — Adverse Event | 0 | 1 | 0
Not completed — Physician Decision | 0 | 1 | 0
Period: PB-102-F02
Arm/Group | 0.2 mg/kg | 1 mg/kg | 2 mg/kg
Started | 6 | 6 | 4
Completed | 6 | 6 | 4
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 0.2 mg/kg | 1 mg/kg | 2 mg/kg | Total
Number analyzed (Participants) | 6 | 8 | 4 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 1 | 0 | 1
  Between 18 and 65 years | 6 | 7 | 4 | 17
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 3 | 7
  Male | 4 | 6 | 1 | 11
Phenotypically Classic vs Non Classic Fabry Patients [Count of Participants; unit: Participants] — Population: A subgroup analysis of patients with phenotypically classic Fabry disease was conducted only in the efficacy group. The efficacy group includes those who completed the study.
  Participants
    number analyzed (Participants) | 6 | 6 | 4 | 16
    Phenotypically Classic Fabry Patients | 5 | 4 | 1 | 10
    Non Classic Fabry Patients | 1 | 2 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: Adverse Events
Description: Reportings of adverse events reported by the patient and from monitoring with clinical laboratory, physical examination and ECG. Results represent the number of AEs that were considered possibly, probably, or definitely related to treatment.
Time Frame: 12 months
Measure: Number; unit: adverse events
Groups:
- Safety Group: The safety population in the study included 18 patients: 6 patients in the 0.2 mg/kg treatment group, 8 patients in the 1.0 mg/kg, and 4 patients in the 2.0 mg/kg treatment groups.
- 1.0 mg/kg: PRX-102 1.0 mg/kg every 2 weeks
- 2.0 mg/kg: PRX-102 2.0 mg/kg every 2 weeks
Arm/Group | Safety Group | 0.2 mg/kg | 1.0 mg/kg | 2.0 mg/kg
Number analyzed (Participants) | 18 | 6 | 8 | 4
adverse events | 54 | 11 | 29 | 14

2. Other Pre Specified Outcome: Plasma Gb3 Concentrations
Description: Results are presented as mean percent change from baseline (visit 1) to 12 months +/- standard error.
Time Frame: Plasma Gb3 concentration (ug/mL) was measured at baseline and every 3 months up to 12 months.
Measure: Mean (Standard Error); unit: mean percent change
Groups:
- Efficacy Group: The efficacy group includes all the subjects that completed the study.
- Phenotypically Classic Fabry Patients: Patients who are phenotypically classic Fabry Patients.
Arm/Group | 0.2 mg/kg | 1 mg/kg | 2 mg/kg | Efficacy Group | Phenotypically Classic Fabry Patients
Number analyzed (Participants) | 6 | 6 | 4 | 16 | 9
mean percent change | -16.8 (8.6) | -30.7 (11.2) | -16.2 (12.7) | -22.2 (6.1) | -33.3 (7.6)

3. Other Pre Specified Outcome: Kidney Function - Change in eGFR
Description: Estimated glomerular filtration rate (eGFR) was calculated by the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation. Levels of eGFR calculated by the CKD-EPI equation, based on measured serum creatinine on day 1, weeks 4, 8, 12, 26, 38 and 52 are used to determine the annualized slope of eGFR per patient over a 12 months period. The absolute mean change from baseline (visit 1) to 12 months is then derived from the eGFR slope.
Time Frame: eGFR is performed at baseline (day 1) weeks 4, 8, 12, 26, 38 and 52 (12 months)
Measure: Mean (Standard Error); unit: mL/min/1.73 m2
Groups:
- Pegunigalsidase Alfa Reporting Group: All 16 patients in the efficacy group, including both phenotypically classic Fabry patients and non classic Fabry patients.
- Phenotypically Classic Fabry Patients: 10 patients who are phenotypically classic Fabry patients.
Arm/Group | Pegunigalsidase Alfa Reporting Group | Phenotypically Classic Fabry Patients
Number analyzed (Participants) | 16 | 10
mL/min/1.73 m2 | -0.8 (1.9) | 0 (2.8)

4. Other Pre Specified Outcome: Plasma Lyso-Gb3 Levels
Description: Results are presented as mean percent change from baseline (visit 1) to 12 months +/- standard error.
Time Frame: Plasma Lyso-Gb3 concentration (ng/mL) was measured at baseline and every 3 months up to 12 months.
Measure: Mean (Standard Error); unit: mean percent change
Arm/Group | 0.2 mg/kg | 1 mg/kg | 2 mg/kg | Efficacy Group | Phenotypically Classic Fabry Patients
Number analyzed (Participants) | 6 | 6 | 4 | 16 | 10
mean percent change | -43.4 (12.2) | -59.9 (7.1) | -40.4 (7.5) | -48.9 (5.7) | -57.6 (6.8)

5. Other Pre Specified Outcome: Change in Kidney Gb3 Accumulation
Description: Kidney biopsy was performed at baseline of study PB-102-F01 and following 6 months treatment with PRX-102. Approximately 300 capillaries were scored in each specimen. A quantitative Barisoni Lipid Inclusion Scoring System (BLISS) was used for scoring Gb3 inclusions in kidney peritubular capillary (PTC) biopsy samples.The scoring system was implemented by 3 blinded pathologists/readers.The BLISS scoring methodology consists of counting the number of Gb-3 inclusions per capillary previously annotated.The final score of each biopsy was the average number of inclusions per capillary. A decrease in scoring from baseline to 6 Month is considered an indication for clinical improvement.
Time Frame: Visit 1 (day 1) in PB-102-F01 study and after a total of 6 months of treatment (i.e., at 3 months into study PB-102-F02).
Population: 3 patients were not included in the renal biopsies Gb3 analysis. 1 male patient's biopsies were mixed up by the lab; 1 female patient's baseline biopsy didn't include cortex tissue making sample unreadable; and 1 male patient carries a cardiac GLA variant (p.N215S) associated with rare renal manifestation and had a low BLISS baseline score
Measure: Mean (Standard Error); unit: Percent change
Arm/Group | Pegunigalsidase Alfa Reporting Group | Phenotypically Classic Fabry Patients
Number analyzed (Participants) | 13 | 8
Percent change | -67.8 (8.9) | -84.1 (3.4)

6. Other Pre Specified Outcome: Cardiac Fibrosis Per MRI
Description: Cardiac MRI was performed to estimate the percentage and mass of the myocardial fibrotic area.
  Results represent the number of subjects with fibrosis after 1 year of treatment.
Time Frame: Cardiac MRI was performed in order to assess myocardial fibrosis at baseline, 6 months and 12 months visit.
Measure: Number; unit: number of subjects
Arm/Group | Pegunigalsidase Alfa Reporting Group | Phenotypically Classic Fabry Patients
Number analyzed (Participants) | 16 | 10
number of subjects | 0 | 0

7. Other Pre Specified Outcome: Cardiac MRI - Ejection Fraction
Description: Results are presented as mean percent change from baseline (visit 1) to 12 months.
Time Frame: Cardiac MRI was performed 3 times: at baseline (visit 1), 6 months and 12 months.
Measure: Mean (Standard Error); unit: Percent Change
Arm/Group | Pegunigalsidase Alfa Reporting Group | Phenotypically Classic Fabry Patients
Number analyzed (Participants) | 16 | 10
Percent Change | -3.1 (3.6) | -7.3 (3.2)

8. Other Pre Specified Outcome: Cardiac MRI - LVM
Description: Results are presented as mean percent change from baseline (visit 1) to 12 months.
Time Frame: Cardiac MRI was performed 3 times: at baseline (visit 1), 6 months and 12 months.
Measure: Mean (Standard Error); unit: Percent change
Arm/Group | Pegunigalsidase Alfa Reporting Group | Phenotypically Classic Fabry Patients
Number analyzed (Participants) | 16 | 10
Percent change | 0 (2.5) | -2.6 (3.4)

9. Other Pre Specified Outcome: Cardiac MRI - LVMI
Description: Cardiac MRI with computer-calculated left ventricular mass index were conducted at baseline, 6 month, and 12 months. Results are presented as mean percent change from baseline (visit 1) to 12 months. LVMI is calculated by dividing the left ventricular mass by body surface area.
Time Frame: Cardiac MRI was performed 3 times: at baseline (visit 1), 6 months and 12 months.
Measure: Mean (Standard Error); unit: Percent Change
Arm/Group | Pegunigalsidase Alfa Reporting Group | Phenotypically Classic Fabry Patients
Number analyzed (Participants) | 16 | 10
Percent Change | 0.4 (2.6) | -3.1 (3.1)

10. Other Pre Specified Outcome: Pharmacokinetics - AUC
Description: PK parameters were derived from the plasma concentration versus time profiles. Results reported represent the averaged values following a single dosing of the study drug.
Time Frame: PK parameters were determined on Day 1 and 3, 6, and 12 months at these time points: pre-infusion (baseline); 1 h after the beginning of the infusion; at the end of the infusion; 1, 4, 8, 24, 48±3, 72±3, 96±3 h and 2 weeks ± 3 days post-infusion.
Measure: Mean (Standard Error); unit: ng*hr/ml
Arm/Group | 0.2 mg/kg | 1 mg/kg | 2 mg/kg
Number analyzed (Participants) | 6 | 6 | 4
ng*hr/ml | 70070 (26044) | 390896 (136476) | 619393 (158562)

11. Other Pre Specified Outcome: Pharmacokinetics - Terminal Half Life
Description: as for outcome 10
Time Frame: as for outcome 10
Measure: Mean (Standard Error); unit: hour
Arm/Group | 0.2 mg/kg | 1 mg/kg | 2 mg/kg
Number analyzed (Participants) | 6 | 6 | 4
hour | 60.3 (19.6) | 78.9 (10.3) | 70.7 (18)

12. Other Pre Specified Outcome: Pharmacokinetics - Clearance of Drug (Cl)
Description: PK parameters were derived from the plasma concentration versus time profiles. Clearance of drug from plasma represents the volume of plasma cleared of the drug per unit time per Kg.
  Results reported represent the averaged values following a single dosing of the study drug.
Time Frame: as for outcome 10
Measure: Mean (Standard Error); unit: ml/hr/kg
Arm/Group | 0.2 mg/kg | 1 mg/kg | 2 mg/kg
Number analyzed (Participants) | 6 | 6 | 4
ml/hr/kg | 2.96 (0.81) | 2.85 (0.66) | 3.41 (0.68)

13. Other Pre Specified Outcome: Pharmacokinetics - Volume of Distribution (Vz)
Description: PK parameters were derived from the plasma concentration versus time profiles. Vz is the volume of distribution during the elimination phase. Results reported represent the averaged values following a single dosing of the study drug.
Time Frame: as for outcome 10
Measure: Mean (Standard Error); unit: ml/kg
Arm/Group | 0.2 mg/kg | 1 mg/kg | 2 mg/kg
Number analyzed (Participants) | 6 | 6 | 4
ml/kg | 246 (68) | 321 (71) | 345 (105)

14. Other Pre Specified Outcome: Pharmacokinetics - Cmax
Description: Pharmacokinetic (PK) parameters were derived from the plasma concentration versus time profiles.
  Cmax is the maximal plasma concentration of a drug after administration. Results reported represent the averaged values following a single dosing of the study drug.
Time Frame: as for outcome 10
Measure: Mean (Standard Error); unit: ng/ml
Arm/Group | 0.2 mg/kg | 1 mg/kg | 2 mg/kg
Number analyzed (Participants) | 6 | 6 | 4
ng/ml | 1858 (531) | 11123 (2409) | 16625 (4299)

15. Other Pre Specified Outcome: Number of Participants With Anti-Drug Antibodies
Description: Results reported represent the number of participants who were tested positive for anti-pegunigalsidase alfa (PRX-102) antibodies, including neutralizing antibodies in patients having a positive IgG antibody response per group, at Visit 1, 2 (Month 1), and then every 2 months during the study, and 2 months after the last infusion.
Time Frame: Anti-pegunigalsidase alfa (PRX-102) antibodies, including neutralizing antibodies in patients having a positive IgG antibody response, were assessed at Visit 1, 2 (Month 1), and then every 2 months during the study, and 2 months after the last infusion.
Measure: Number; unit: participants
Arm/Group | 0.2 mg/kg | 1 mg/kg | 2 mg/kg | Efficacy Group
Number analyzed (Participants) | 6 | 6 | 4 | 16
participants | 2 | 1 | 0 | 3

16. Other Pre Specified Outcome: Change in Short Form Brief Pain Inventory (BPI)
Description: Pain severity (worst, least, average, and right now) is summarized at baseline, 3-month, 6-month and 12-month of the study. The Short Form Brief Pain Inventory (BPI) is based on a 10-point scale, where 0=no pain and 10=pain as bad as you can imagine. A reduction in pain severity score indicated an improvement. The changes from baseline for individual scores and composite scores (a mean severity score) was assessed. The mean change in score from baseline at the 12-month visit is reflected.
Time Frame: The Short Form Brief Pain Inventory (BPI) is assessed at baseline, 3-month, 6-month, and 12-month visits.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Pegunigalsidase Alfa Reporting Group | Phenotypically Classic Fabry Patients
Number analyzed (Participants) | 16 | 10
score on a scale | -0.7 (0.4) | -1.2 (0.4)

17. Other Pre Specified Outcome: Urine Creatinine Level
Description: Proteinuria is assessed using spot urine tests at baseline, 3-month, 6-month, 9-month, and 12-month visits. The percent changes of urine creatinine level at the 12-month visit from baseline is reflected.
Time Frame: Urine creatinine level is assessed at baseline, 3-month, 6-month, 9-month, and 12-month visits using spot urine tests.
Measure: Mean (Standard Error); unit: Percentage change from baseline
Arm/Group | 0.2 mg/kg | 1 mg/kg | 2 mg/kg | Efficacy Group
Number analyzed (Participants) | 6 | 6 | 4 | 16
Percentage change from baseline | -15.9 (25.6) | -15.3 (27.8) | -68.3 (2.5) | -28.8 (14.6)

18. Other Pre Specified Outcome: Urine Protein/Creatinine Ratio
Description: Proteinuria is assessed using spot urine tests at baseline, 3-month, 6-month, 9-month, and 12-month visits. The percent changes of urine protein/creatinine ratio at the 12-month visit from baseline is reflected.
Time Frame: Protein/.creatinine ratio is assessed at baseline, 3-month, 6-month, 9-month, and 12-month visits
Measure: Mean (Standard Error); unit: Percentage change from baseline
Arm/Group | 0.2 mg/kg | 1 mg/kg | 2 mg/kg | Efficacy Group
Number analyzed (Participants) | 6 | 6 | 4 | 16
Percentage change from baseline | -2.6 (23.4) | -14.8 (14.1) | -7.9 (12.4) | -8.5 (10.1)

19. Other Pre Specified Outcome: Total Urine Protein Level
Description: Proteinuria is assessed using spot urine tests at baseline, 3-month, 6-month, 9-month, and 12-month visits. The percent changes of total urine protein level at the 12-month visit from baseline is reflected.
Time Frame: Total urine protein level is assessed at baseline, 3-month, 6-month, 9-month, and 12-month visits.
Measure: Mean (Standard Error); unit: Percentage change from baseline
Arm/Group | 0.2 mg/kg | 1 mg/kg | 2 mg/kg | Efficacy Group
Number analyzed (Participants) | 6 | 6 | 4 | 16
Percentage change from baseline | -35.1 (18.4) | -32.8 (17.4) | -71.7 (7.3) | -43.4 (9.9)

20. Other Pre Specified Outcome: Brain MRI
Description: Qualitative assessments regarding evidence of stroke using brain MRI were summarized at baseline and 12-month visits. Number is subjects with evidence of stoke on the brain MRI at the 12-month visit is reflected.
Time Frame: Brain MRI is performed at baseline and 12-month visit.
Measure: Count of Participants; unit: Participants
Arm/Group | 0.2 mg/kg | 1 mg/kg | 2 mg/kg | Efficacy Group
Number analyzed (Participants) | 6 | 6 | 4 | 16
Participants | 0 | 0 | 0 | 0

21. Other Pre Specified Outcome: Change in Mainz Severity Score Index (MSSI)
Description: The Mainz Severity Score Index (MSSI) is useful for monitoring clinical improvement in patients receiving enzyme replacement therapy. The MSSI scoring system is composed of four sections that cover the general, neurological,cardiovascular and renal signs and symptoms of Fabry disease. Each section includes a group of signs and symptoms that are associated with Fabry disease. The minimal score is 0, and the maximum score for the general section is 18. A higher score indicates more severe clinical manifestations of the disease.The MSSI is performed at baseline, 6-month, and 12-month. The overall mean reduction of the total general score at 12-month from baseline is reflected.
Time Frame: The MSSI is performed at baseline, 6-month, and 12-month
Measure: Mean (Standard Error); unit: score of a scale
Arm/Group | 0.2 mg/kg | 1 mg/kg | 2 mg/kg | Efficacy Group
Number analyzed (Participants) | 6 | 6 | 4 | 16
score of a scale | -2.8 (1.2) | -1.2 (0.6) | -1.5 (0.9) | -1.9 (0.6)

22. Other Pre Specified Outcome: Gastrointestinal Symptoms Questionnaire - Severity of Abdominal Pain
Description: A qualitative assessments regarding abdominal pain and diarrhea at baseline, 3-month, 6-month, 9-month, and 12-month visits. The subjects were asked to report the severity of their abdominal pain as no pain, mild, moderate, severe or really severe. The number of subjects who reported no or mild abdominal pain at the 12-month visit are reflected.
Time Frame: The Gastrointestinal Symptoms Questionnaire is assessed at baseline, 3-month, 6-month, 9-month, and 12-month visits.
Measure: Number; unit: participants
Arm/Group | Pegunigalsidase Alfa Reporting Group | Phenotypically Classic Fabry Patients
Number analyzed (Participants) | 16 | 10
participants | 10 | 7

23. Other Pre Specified Outcome: Gastrointestinal Symptoms Questionnaire - Frequency of Abdominal Pain
Description: A qualitative assessments regarding abdominal pain and diarrhea at baseline, 3-month, 6-month, 9-month, and 12-month visits. The subjects were asked to report their frequency of abdominal pain as never, rarely, monthly, weekly, or daily. The numbers of subjects who reported never or rarely having abdominal pain at the 12-month visit are reflected.
Time Frame: The Gastrointestinal Symptoms Questionnaire is assessed at baseline, 3-month, 6-month, 9-month, and 12-month visits.
Measure: Count of Participants; unit: Participants
Arm/Group | Pegunigalsidase Alfa Reporting Group | Phenotypically Classic Fabry Patients
Number analyzed (Participants) | 16 | 10
Participants | 7 | 5

24. Other Pre Specified Outcome: Gastrointestinal Symptoms Questionnaire - Frequency of Diarrhea
Description: A qualitative assessments regarding abdominal pain and diarrhea at baseline, 3-month, 6-month, 9-month, and 12-month visits. The subjects were asked to report their frequency of diarrhea as never, rarely, monthly, weekly, or daily. The number of subjects who reported never or rarely having diarrhea at the 12-month visit is reflected.
Time Frame: The Gastrointestinal Symptoms Questionnaire is assessed at baseline, 3-month, 6-month, 9-month, and 12-month visits.
Measure: Count of Participants; unit: Participants
Arm/Group | Pegunigalsidase Alfa Reporting Group | Phenotypically Classic Fabry Patients
Number analyzed (Participants) | 16 | 10
Participants | 11 | 6

ADVERSE EVENTS:
Time Frame: AEs were collected from the start of treatment throughout the 12 months of the study, plus a follow-up visit 2 months after 12-months study visit.
Groups:
- 1 mg/kg: PRX-102 1.0 mg/kg every 2 weeks
- 2 mg/kg: PRX-102 2.0 mg/kg every 2 weeks
Arm/Group | 0.2 mg/kg | 1 mg/kg | 2 mg/kg
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/8 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/6 | 1/8 | 1/4
Other Adverse Events (participants affected / at risk) | 2/6 | 7/8 | 2/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 0.2 mg/kg (N=6) | 1 mg/kg (N=8) | 2 mg/kg (N=4)
Renal Hematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0 — One patient in the 1mg/kg group experienced a renal hematoma due to the kidney biopsy at baseline. The patient was treated and the renal hematoma was resolved. This event was considered unrelated to treatment.
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 — A 52 y.o. male experienced a bronchospasm related to the study drug 40 minutes following the first infusion initiation, was treated, recovered, and discontinued Per Protocol. Anti PRX-102 IgG was negative and anti PRX-102 IgE was positive at baseline
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 0.2 mg/kg (N=6) | 1 mg/kg (N=8) | 2 mg/kg (N=4)
Hypotension (Vascular disorders) | 0 (0) | 1 (3) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Chest pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (3) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Chest discomfort (General disorders) | 1 (2) | 1 (1) | 0 (0)
Infusion reaction (General disorders) | 0 (0) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (2) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (7)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0)
Itching (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Sweating (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0)
Corneal Edema (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Conjunctival Hemorrhage (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Edema (General disorders) | 1 (1) | 0 (0) | 0 (0)
Peripheral Edema (General disorders) | 1 (1) | 0 (0) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Visual field defect (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Typical aura without headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2)
Fatigue (General disorders) | 0 (0) | 2 (6) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal Stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Nervousness (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes